CLINICAL TRIAL: NCT01765985
Title: Treatment of Palmoplantar Psoriasis With Low Doses Interferential Current
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pr PASSERON (Other)
Responsible Party: Sponsor-Investigator, Pr PASSERON, Professor, Association Niçoise Pour la Recherche En Dermatologie
Organization: Association Niçoise Pour la Recherche En Dermatologie (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-CRO-01
Record Dates: First submitted 2012-12-06; First posted 2013-01-11 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Psoriasis Palm & Soles
Keywords: palmoplantar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intercurrent PSORIAMED (Experimental): 5 minutes twice a day for 12 weeks
  Interventions: Device: PSORIAMED
- PLACEBO (Active Comparator): V0 : Selection: Information of the patient, control of inclusion and non inclusion criteria.
  V1 : Control of inclusion and non inclusion criteria (treatment against psoriasis have to be discontinued for at least 3 weeks and 3 months for anti-IL12/23). Clinical scores and photographs. Explanation of the functioning of the device, then the treatment is followed at home, twice a day 5 minutes. 10% salicylic acid ointment will be applied after each session.
  V2 : End of the treatment (12 weeks after V1). Clinical scores and photographs. V3 : End of the follow-up (24 weeks after V1). Clinical scores and photographs.
  Interventions: Device: PLACEBO

INTERVENTIONS:
Device: PSORIAMED — V0 : Selection: Information of the patient, control of inclusion and non inclusion criteria.
  V1 : Control of inclusion and non inclusion criteria (treatment against psoriasis have to be discontinued for at least 3 weeks and 3 months for anti-IL12/23). Clinical scores and photographs. Explanation of the functioning of the device, then the treatment is followed at home, twice a day 5 minutes. 10% salicylic acid ointment will be applied after each session.
  V2 : End of the treatment (12 weeks after V1). Clinical scores and photographs. V3 : End of the follow-up (24 weeks after V1). Clinical scores and photographs.
  Arms: Intercurrent PSORIAMED
Device: PLACEBO — V0 : Selection: Information of the patient, control of inclusion and non inclusion criteria.
  V1 : Control of inclusion and non inclusion criteria (treatment against psoriasis have to be discontinued for at least 3 weeks and 3 months for anti-IL12/23). Clinical scores and photographs. Explanation of the functioning of the device, then the treatment is followed at home, twice a day 5 minutes. 10% salicylic acid ointment will be applied after each session.
  V2 : End of the treatment (12 weeks after V1). Clinical scores and photographs. V3 : End of the follow-up (24 weeks after V1). Clinical scores and photographs.
  Arms: PLACEBO

SUMMARY:
Interferential current has shown promising results for treating psoriasis with a good tolerance. Prospective randomized studies versus placebo are required to confirm the interest of such an approach.

The Main objective is to assess the efficacy of interferential current for treating palmoplantar psoriasis.

Secondary objectives is to assess the subjective efficacy by the patients, the efficacy on the nails, to study the potential side effects.

DETAILED DESCRIPTION:
Interferential current has shown promising results for treating psoriasis with a good tolerance. Prospective randomized studies versus placebo are required to confirm the interest of such an approach.

Main objective To assess the efficacy of interferential current for treating palmoplantar psoriasis.

Secondary objectives To assess the subjective efficacy by the patients, the efficacy on the nails, to study the potential side effects.

Patients Patients from 18 to 90 year-old with psoriasis on the hands and/or feet. Length of the study: 12 months Methods Monocentric randomized comparative study versus placebo.Intervention V0 : Selection: Information of the patient, control of inclusion and non inclusion criteria.

V1 : Control of inclusion and non inclusion criteria (treatment against psoriasis have to be discontinued for at least 3 weeks and 3 months for anti-IL12/23). Clinical scores and photographs. Explanation of the functioning of the device, then the treatment is followed at home, twice a day 5 minutes. 10% salicylic acid ointment will be applied after each session.

V2 : End of the treatment (12 weeks after V1). Clinical scores and photographs. V3 : End of the follow-up (24 weeks after V1). Clinical scores and photographs.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 90 year-old with psoriasis on the hands and/or feet diagnosed clinically

Exclusion Criteria:

* Pregnant women,
* implantable electronic device (such as pace maker), betabloquer.
* Concomitant use of a treatment potentially active on psoriasis (steroids, vitamin D analogues, immunosuppressive drug, acitretin, cyclosporine, methotrexate, anti-TNF, anti-IL12/IL23).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Test IGA | 12 weeks
  IGA (investigator Global assessment) score from 0 (healed) to 4 (worst) at 12 and 24 weeks. The criteria of success will be IGA 0 or 1 at W12.

SECONDARY OUTCOMES:
PASI (Psoriasis Activity Severity Index) | 12 weeks
  PASI (Psoriasis Activity Severity Index)
PGA (Patient global assessment) | 12 weeks
  PGA (Patient global assessment)
NAPSI (Nail Activity Psoriasis Severity Index) | 12 weeks
  NAPSI (Nail Activity Psoriasis Severity Index)

CONTACTS AND LOCATIONS:
Overall Officials: PASSERON Thierry, Pu-Ph, Principal Investigator — ANPRED - Service de Dermatologie - Hôpital de l'Archet - 151 Route de saint-antoine de ginestière 06200 Nice
Locations (1):
- ANPRED - Hôpital de l'archet - 151 route de sainte antoine de ginestière, Nice, Alpes-Maritimes, France